CLINICAL TRIAL: NCT02292680
Title: Novel Biomarkers for Exposures in the Neonatal Intensive Care Unit
Brief Title: Childhood Measures of NICU-based Chemical Exposure
Status: Withdrawn | Type: Observational
Why Stopped: Unable to enroll
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 14-1403
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Development
Keywords: dentin; environmental exposures; neurodevelopmental outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- NICU Tooth Study Cohort: All study subjects will have been cared for in the Mount Sinai NICU and have had the same hospital environment exposure.

SUMMARY:
This study aims to identify early life exposures to metals and chemicals by measuring the concentration of metals and organic compounds in shed primary teeth. The researchers will also investigate associations between the presence of these chemicals in teeth and children's social, emotional, and neuro-development.

DETAILED DESCRIPTION:
Since children begin shedding their primary teeth around age 6, the investigators will enroll children who will be turning 6 in the next two years. First, the investigators will follow up with the children's development by conducting a battery of non-invasive neurodevelopmental tests. Also, the parents will be asked to complete a questionnaire called the Child Behavior Checklist, which assesses behavioral problems. Then, each child's parent will be asked to send the research team 2-3 teeth that their child has shed, or to send teeth as they are shed over the next three years. Dr. Stroustrup's collaborator, Dr. Manish Arora, will perform a temporal analysis of chemical distribution for each tooth to determine each child's environmental exposures during the perinatal and neonatal periods.

ELIGIBILITY:
Inclusion Criteria:

* 4-6 years of age in 2014 (six years of age by the end of 2016)
* Cared for as a neonate in Mount Sinai's NICU

Exclusion Criteria:

* Parent documented in Mount Sinai's database is no longer the legal guardian
* Non-English-speaking parents

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children who were cared for as neonates in the Mount Sinai NICU
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01 (Estimated); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Chemical Concentration in deciduous teeth | up to 5 years
  Teeth will be analyzed by a dentist and researcher trained in laser ablation inductively coupled plasma mass spectroscopy technology

SECONDARY OUTCOMES:
Child Behavior Checklist | up to 3 years
  An assessment Developmental Outcomes measured using this assessments
Wechsler Preschool and Primary Scale of Intelligence | up to 3 years
  Developmental Outcomes measured using this assessments
Development Neuropsychological Assessment (NEPSY) | up to 3 years
  Developmental Outcomes measured using this assessments

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie Stroustrup, MD,MPH, Principal Investigator — Ichan School of Medicine at Mount Sinai